CLINICAL TRIAL: NCT02408458
Title: A Prospective Post-Market Clinical Evaluation of Miromatrix Biological Mesh for Ventral Hernia Repair
Brief Title: Miromatrix Biological Mesh for Ventral Hernia Repair
Acronym: MIROMESH PM-1
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment rate
Sponsor: Miromatrix Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015001
Record Dates: First submitted 2015-03-26; First posted 2015-04-03 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-10

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MIROMESH (Other): Single-arm study. MIROMESH will be used in the surgical repair of ventral hernia.
  Interventions: Device: MIROMESH®

INTERVENTIONS:
Device: MIROMESH®

SUMMARY:
This study is being conducted to gather long-term data of the performance of the Miromatrix Biological Mesh.

DETAILED DESCRIPTION:
Miromatrix Medical Inc. has developed a new biologic mesh, called MIROMESH®. MIROMESH received FDA 510(k) clearance with an indication for reinforcement of soft tissue on March 31, 2014 under K134033. Miromatrix Biologic Mesh is a non cross-linked, acellular surgical mesh that is derived from the highly vascularized porcine liver. This study will serve to provide clinicians with high-quality clinical data in order to provide them with a higher degree of confidence when selecting MIROMESH for ventral hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 80 years old on the day of study enrollment
* ventral or incisional hernia greater than 9 cm2 for which the physician anticipates ability to achieve midline fascia closure following a retro-rectus repair/component separation
* hernia classified as CDC class 1 or 2 preoperatively
* able and willing to sign the consent form and comply with all study visits and procedures
* commit to non-smoking for at least 4 weeks prior to procedure

Exclusion Criteria:

* sensitivity to porcine material
* scheduled for a concomitant procedure of a wound classified as other than clean
* immunocompromised or at risk of immunosuppression (i.e. be HIV positive, be experiencing organ rejection, be a recent or anticipated chemotherapy recipient) as determined by the Investigator
* BMI ≥40
* A1C level ≥10.0
* participating in another clinical study
* cirrhosis, and/or ascites
* diagnosed with a collagen vascular disorder
* American Society of Anesthesiology (ASA) Class 4 or 5
* allergic to tetracycline or kanacmycin
* life expectancy of less than 2 years at the time of enrollment
* any condition in the opinion of the Investigator that would preclude the use of the study device, or preclude the subject from completing the follow-up requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Hernia recurrence requiring surgical intervention | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: J. Scott Roth, M.D., Principal Investigator — University of Kentucky
Locations (4):
- United States (4):
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University of Kentucky, Lexington, Kentucky
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin